CLINICAL TRIAL: NCT07178379
Title: HARP Trial: Hysteroscopy Anesthesia for Relief of Pain
Brief Title: Hysteroscopy Anesthesia for Relief of Pain
Acronym: HARP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Principal Investigator, Paula Caballero, MD Obstetrics and Gynecology Reina Sofia Hospital, Maimónides Biomedical Research Institute of Córdoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HARP
Record Dates: First submitted 2025-08-02; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Pain Management; Outpatient Hysteroscopy; Local Anesthesia; Procedural Pain Relief; Gynecologic Procedure
Keywords: hysteroscoy; outpatient hysteroscopy; pain assessment; visual analog scale; localanesthesia; ambulatory surgery; randomized controlled trial
MeSH Terms: conditions — Agnosia | interventions — Anesthesia, Local; Mepivacaine

STUDY DESIGN:
Who Masked: Participant
Masking Description: This is a single-blind study with partial masking. Patients will not be explicitly informed whether they are receiving local anesthesia or placebo. In the control group, a simulated intervention (saline irrigation of the cervix and vagina) will be performed to mimic the anesthetic procedure. However, due to the nature of the intervention (injection of anesthetic vs. no injection), full blinding of patients is not feasible.
  The healthcare provider administering the intervention is not blinded, but both the principal investigator and the statistician will be blinded to group allocation during data analysis. This aims to reduce observer and analysis bias
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Patients in the control group will undergo a placebo-like intervention in which the vagina and cervix will be irrigated with 0.9% normal saline using a syringe, simulating the motion and timing of the anesthetic application without actual injection. This aims to reduce expectation bias. No active anesthetic agent will be used.
  Intervention Type: Placebo Comparator Substance: Saline (0.9% sodium chloride) Route: Vaginal and cervical irrigation Purpose: To serve as the control arm for comparison of pain levels in patients not receiving anesthetic injections.
  Interventions: Other: Placebo
- Local Anesthesia (Mepivacaine 3%) (Experimental): Patients in this group will receive an injection of 3% mepivacaine into the uterosacral ligaments before undergoing diagnostic hysteroscopy. The anesthetic will be administered using a 25 mm Carpule needle, with 3.4 mL injected into each uterosacral ligament under standard gynecological positioning. The procedure will begin approximately one minute after administration to allow time for the anesthetic effect.
  Intervention Type: Drug Drug Name: Mepivacaine 3% Dose and Route: Local injection - 6.8 mL total (3.4 mL per side) Purpose: To assess the effect of local anesthesia on pain perception during outpatient hysteroscopy.
  Interventions: Procedure: Local paracervical Anesthesia

INTERVENTIONS:
Procedure: Local paracervical Anesthesia — 1. Intervention Group (Local Anesthesia) Name: Mepivacaine 3% uterosacral ligament block Type: Pharmacological (local anesthetic).
  Dose/Administration:
  Drug: Mepivacaine hydrochloride 3% (4 vials of 1.7 mL each, total 6.8 mL). Route: Bilateral injection into uterosacral ligaments (2 injections per ligament, 3.4 mL per side).
  Technique:
  Patient in lithotomy position. Uterosacral ligaments identified posteriorly to the cervix. Injection with a 27G Carpule needle (25 mm length) at 2-3 mm depth. Slow infusion (to minimize dispersion). Timing: Administered ≥1 minute before hysteroscopy.
  Other Names: local anesthesia; mepivacaine; Mepivacaine 3% uterosacral ligament block
  Arms: Local Anesthesia (Mepivacaine 3%)
Other: Placebo — Procedure:
  Vaginal and cervical irrigation with 0.9% saline solution (4 irrigations, mimicking anesthesia administration).
  Mimicry:
  Same equipment (syringe, speculum) as intervention group. Identical patient positioning and timing
  Other Names: Saline irrigation (sham procedure); Non-pharmacological
  Arms: Control

SUMMARY:
This randomized clinical trial aims to evaluate the effect of local anesthesia on pain perception in patients undergoing outpatient diagnostic hysteroscopy. Although generally well tolerated, pain during hysteroscopy remains a leading cause of procedural failure and patient discomfort. Current evidence on the effectiveness of local anesthetic techniques is limited, with considerable variability in study designs, patient populations, and outcomes measured.

This study will compare pain levels between two groups: one receiving local anesthetic infiltration (3% mepivacaine into the uterosacral ligaments), and the other undergoing a placebo-like intervention (saline irrigation without injection). Pain will be assessed using a standardized Visual Analog Scale (VAS).

The primary objective is to determine whether local anesthesia significantly reduces pain perception during the procedure. Secondary objectives include evaluating which patient or procedural variables may influence pain (e.g., parity, uterine position, BMI, operator experience) and whether local anesthesia impacts the need for post-procedural analgesia or complication rates.

Patients will be randomly assigned in a 1:1 ratio using a simple randomization method. Although the study design does not allow for double blinding, efforts will be made to minimize expectation bias-patients will not be explicitly informed whether they are receiving anesthesia or not, and the placebo group will receive simulated intervention. The principal investigator and the statistician will be blinded to the treatment allocation during data analysis.

Inclusion criteria are: age ≥ 18 years, indication for office-based diagnostic hysteroscopy or minor operative procedures (e.g., polypectomy or biopsy), and no previous hysteroscopy experience. Exclusion criteria include known anesthetic allergy, complex procedures (e.g., myomectomy), anatomic uterine malformations, severe complications, or lack of consent.

A total sample size of 58 patients (29 per group) has been calculated based on an expected clinically relevant VAS difference of 1.5 points and a standard deviation of 2.0. To account for possible dropouts, up to 70 patients may be enrolled.

The results of this trial will provide higher quality evidence on whether local anesthesia should be routinely recommended in outpatient hysteroscopy and may support cost-effectiveness studies in the future.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years: To ensure that participants are legal adults and able to provide informed consent.
* Indication for office-based diagnostic hysteroscopy: The patient must be scheduled for a diagnostic hysteroscopy, either for uterine cavity evaluation or diagnostic purposes.
* Simple procedures like uterine polypectomies involving 1, 2, or more than 3 polyps or endometrial biopsy
* No previous hysteroscopies

Exclusion Criteria

* Age < 18 years
* Known allergy to any local anesthetic
* General contraindications to hysteroscopy including pregnancy (established via interview, last menstrual period, contraceptive use, or pregnancy test), active infection (e.g., pyometra or recent pelvic inflammatory disease), recent uterine perforation, etc.
* Complex procedures like myomectomy with morcellator
* Failure to access the uterine cavity
* Anatomic conditions preventing cavity access
* Excessive procedure duration or fluid use (fluid deficit > 1000 cc)
* Known uterine malformations
* Waiting times exceeding 60 minutes
* Use of analgesic medication prior to the procedure
* Major complications related to the procedure including uterine perforation, creation of a false passage, or significant bleeding requiring interventions beyond standard care.
* Incomplete delivery of informed consent or failure to complete the pre-procedure anxiety questionnaire.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2025-09-06 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity during hysteroscopy | Immediately after the procedure
  Pain will be measured using a 10-point Visual Analog Scale (VAS) immediately after the procedure. Patients will be asked to rate the maximum pain experienced during the hysteroscopy.
  Measure Type: Continuous (VAS score 0-10) Unit of Measure: Points on VAS scale Method of Aggregation: Mean (± SD) Statistical Analysis Plan: Comparison between groups using Student's t-test or Mann-Whitney U test depending on normality.

SECONDARY OUTCOMES:
Need for post-procedure analgesia | Within 30 minutes post-procedure
  Whether patients required any analgesic medication after the hysteroscopy, and what type.
  Measure Type: Binary (Yes/No), plus qualitative record of analgesic used Unit of Measure: Proportion of patients (%)
Procedure-related complications | During and immediately after the procedure
  Description:
  Recording of any intraoperative or immediate postoperative complications (e.g., vasovagal episodes, perforation, bleeding).
  Measure Type: Binary (Yes/No), with qualitative subtype Unit of Measure: Number of events
Indication for surgical hysteroscopy due to intolerable pain | Immediately post-procedure
  Description:
  Whether the patient had to be referred for surgical hysteroscopy under anesthesia due to failure or intolerance of office hysteroscopy.
  Measure Type: Binary (Yes/No) Unit of Measure: Number of cases

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Garcia Fernandez, MD, Principal Investigator, Principal Investigator — MD Obstetrics and Gynecology Reina Sofia Hospital, Cordoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Al-Sunaidi M, Tulandi T. A randomized trial comparing local intracervical and combined local and paracervical anesthesia in outpatient hysteroscopy. J Minim Invasive Gynecol. 2007 Mar-Apr;14(2):153-5. doi: 10.1016/j.jmig.2006.09.007. PMID 17368248
- [Result] Kokanali MK, Guzel AI, Ozer I, Topcu HO, Cavkaytar S, Doganay M. Pain experienced during and after office hysteroscopy with and without intracervical anesthesia. J Exp Ther Oncol. 2014;10(4):243-6. PMID 25509976
- [Result] Vercellini P, Colombo A, Mauro F, Oldani S, Bramante T, Crosignani PG. Paracervical anesthesia for outpatient hysteroscopy. Fertil Steril. 1994 Nov;62(5):1083-5. PMID 7646610
- [Result] Cooper NA, Khan KS, Clark TJ. Local anaesthesia for pain control during outpatient hysteroscopy: systematic review and meta-analysis. BMJ. 2010 Mar 23;340:c1130. doi: 10.1136/bmj.c1130. PMID 20332307
- [Result] Ahmad G, Saluja S, O'Flynn H, Sorrentino A, Leach D, Watson A. Pain relief for outpatient hysteroscopy. Cochrane Database Syst Rev. 2017 Oct 5;(10)(10):CD007710. doi: 10.1002/14651858.CD007710.pub3. PMID 35611933
- [Result] De Silva PM, Carnegy A, Smith PP, Clark TJ. Local anaesthesia for office hysteroscopy: A systematic review & meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2020 Sep;252:70-81. doi: 10.1016/j.ejogrb.2020.05.062. Epub 2020 Jun 2. PMID 32570188
- [Result] Huang L, Yu Q, Zhu Z, Huang P, Ding X, Ma X, Chen Y, Su D. The Current Situation of Anaesthesia for Hysteroscopy in Mainland China: A National Survey. J Pers Med. 2023 Sep 26;13(10):1436. doi: 10.3390/jpm13101436. PMID 37888047
- [Result] Nowak A, Chmaj-Wierzchowska K, Lach A, Malinger A, Wilczak M. Evaluation of Pain During Hysteroscopy Under Local Anesthesia, Including the Stages of the Procedure. J Clin Med. 2024 Nov 21;13(23):7030. doi: 10.3390/jcm13237030. PMID 39685488

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-09-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT07178379/Prot_ICF_000.pdf